CLINICAL TRIAL: NCT05528770
Title: Evaluation of The Postprandial Impact of Automated Priming Bolus for Full Closed Loop Insulin Delivery
Acronym: Rocket-BPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marc Breton (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Marc Breton, Associate Director for Research, Center for Diabetes Technology, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 220261; R01DK129553 (NIH)
Record Dates: First submitted 2022-08-29; First posted 2022-09-06 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes
Keywords: Continuous Glucose Monitor (CGM); Continuous subcutaneous insulin infusion (CSII); Closed Loop Control (CLC); Hybrid Closed Loop (HCL); High-intensity interval training (HIIT); Bolus Priming System (BPS); Fully Automated Closed Loop (FCL); Artificial Pancreas (AP)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the order that they experience the use of the Bolus Priming System (BPS) in fully automated closed loop (FCL) (for 24 hours each, with a 24-hour challenge period in between): 1) with the BPS active, 2) BPS inactive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Full closed-loop (FCL) with Bolus Priming System (BPS) followed by FCL without BPS (Active Comparator): Two separate 24-hour periods during where fully closed loop (FCL) control is used with & without the Bolus Priming system (BPS) active (BPS is designed to recognize meal ingestion & deliver a quick priming dose of insulin prior to extreme blood sugar excursions.) These will be separated by a 24-hour challenge period which will involve further meal & exercise challenges. During these 24-hour periods, participants will be followed for the experimental meals as part of the Study Controller Sessions to compare blood glucose control with & without the BPS. The study meals & activities will be standardized between study sessions.
  During a washout period, we will test the RocketAP system in FCL with further challenges:
  * A session of high-intensity interval training
  * A high-carbohydrate, high-fat meal
  * Ingestion of a bolus of simple sugar
  Interventions: Device: FCL+BPS; Device: FCL
- Full closed-loop (FCL) without Bolus Priming System (BPS) followed by FCL with BPS (Active Comparator): Two separate 24-hour periods during where fully closed loop (FCL) control is used with & without the Bolus Priming system (BPS) active (BPS is designed to recognize meal ingestion & deliver a quick priming dose of insulin prior to extreme blood sugar excursions.) These will be separated by a 24-hour challenge period which will involve further meal & exercise challenges. During these 24-hour periods, participants will be followed for the experimental meals as part of the Study Controller Sessions to compare blood glucose control with & without the BPS. The study meals & activities will be standardized between study sessions.
  During a washout period, we will test the RocketAP system in FCL with further challenges:
  * A session of high-intensity interval training
  * A high-carbohydrate, high-fat meal
  * Ingestion of a bolus of simple sugar
  Interventions: Device: FCL+BPS; Device: FCL

INTERVENTIONS:
Device: FCL+BPS — The automated insulin delivery system includes the Bolus Priming System, a software automatically analyzing past continuous glucose monitoring values to trigger priming insulin bolus delivery isn the suspected presence of meal like glycemic disturbances
  Other Names: Full closed-loop (FCL) with Bolus Priming System
Device: FCL — The automated insulin delivery system does not include the Bolus Priming System, and therefore does not automatically command priming boluses.
  Other Names: Full closed-loop (FCL) without Bolus Priming System

SUMMARY:
The purpose of this study is to understand the impact of the automated priming boluses on the safety and feasibility of a new fully automated AP controller.

DETAILED DESCRIPTION:
Study participants will be admitted to the hotel for a 4-night study, receiving the two sessions in random order: 1) Fully control loop (FCL) with the bolus priming system (BPS) activated, 2) FCL without the BPS, with a 24-hour washout period in between. During the admission, participants will receive structured meals and have blood glucose control followed to compare time in range 70-180 mg/dL between Controller sessions. After the first 24 hour period on the first FCL approach (BPS vs. no BPS,) that the participant has been randomized to, there will be a 24 hour challenge period before shifting to the other randomized approach; during this session participants will undergo further testing of the control algorithm, including meal challenges and a high-intensity interval training bout.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.0 and ≤65 years old at time of consent
2. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year
3. Currently using insulin for at least six months
4. Currently using insulin pump for at least three months
5. Using insulin parameters such as carbohydrate ratio and correction factors consistently on their pump in order to dose insulin for meals or corrections
6. Current regular exercise (e.g. walk, bike, jog) and be able to participate in a high intensity interval training activity.
7. Access to internet and willingness to upload data during the study as needed
8. For females, not currently known to be pregnant or breastfeeding
9. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
10. Willingness to suspend use of any personal CGM for the duration of the clinical trial once the study CGM is in use
11. Willingness to use the UVa closed-loop system throughout study admission
12. Willingness to use personal lispro (Humalog) or aspart (Novolog) during the study admission.
13. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial (including metformin/biguanides, GLP-1 receptor agonists, pramlintide, DPP-4 inhibitors, sulfonylureas and naturaceuticals)
14. Willingness to eat at least 1 g/kg of carbohydrate per day during the hotel admission
15. Willingness to reschedule if placed on oral steroids
16. An understanding and willingness to follow the protocol and signed informed consent
17. Willingness to follow COVID-19 protocols in place at the time of study.

Exclusion Criteria:

1. History of diabetic ketoacidosis (DKA) in the 6 months prior to enrollment
2. Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
3. Pregnancy or intent to become pregnant during the trial
4. Currently being treated for a seizure disorder
5. Planned surgery during study duration.
6. Treatment with meglitinides/sulfonylureas at the time of hotel study.
7. Use of metformin/biguanides, GLP-1 agonists, pramlintide, DPP-4 inhibitors, SGLT-2 inhibitors, or naturaceuticals with a change in dose in the past month.
8. Coronary artery disease or heart failure, unless written clearance is received from a cardiologist or personal health care provider allowing clearance for high-intensity interval training and documentation of a negative stress test within the year
9. History of cardiac arrhythmia (except for benign premature atrial contractions and benign premature ventricular contractions which are permitted or previous ablation of arrhythmia without recurrence which may be permitted)
10. Clinically significant electrocardiogram (ECG) at time of Screening, as interpreted by the study medical physician.
11. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

    1. Inpatient psychiatric treatment in the past 6 months
    2. Presence of a known adrenal disorder
    3. Abnormal liver function test results (Transaminase >2 times the upper limit of normal); testing required for subjects taking medications known to affect liver function or with diseases known to affect liver function
    4. Uncontrolled thyroid disease
    5. Musculoskeletal or other condition that limits participation in exercise portion of study
12. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol.
13. Positive Covid-19 test result

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Brown, MD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Moscoso-Vasquez M, Colmegna P, Barnett C, Fuller M, Koravi CLK, Brown SA, DeBoer MD, Breton MD. Evaluation of an Automated Priming Bolus for Improving Prandial Glucose Control in Full Closed Loop Delivery. Diabetes Technol Ther. 2025 Feb;27(2):93-100. doi: 10.1089/dia.2024.0315. Epub 2024 Nov 6. PMID 39501832

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 participants signed informed consent for the main study. 2 screen failed and 2 withdrew prior to randomization to arms. Results reported on 11 participants who were randomized.
Groups:
- Full Closed-loop (FCL) With Bolus Priming System (BPS) Followed by FCL Without BPS; Full Closed-loop (FCL) Without Bolus Priming System (BPS) Followed by FCL With BPS: Two separate 24-hour periods during where fully closed loop (FCL) control is used with & without the Bolus Priming system (BPS) active (BPS is designed to recognize meal ingestion & deliver a quick priming dose of insulin prior to extreme blood sugar excursions.) These will be separated by a 24-hour challenge period which will involve further meal & exercise challenges. During these 24-hour periods, participants will be followed for the experimental meals as part of the Study Controller Sessions to compare blood glucose control with & without the BPS. The study meals & activities will be standardized between study sessions.
  During a washout period, we will test the RocketAP system in FCL with further challenges:
  * A session of high-intensity interval training
  * A high-carbohydrate, high-fat meal
  * Ingestion of a bolus of simple sugar
  FCL+BPS: The automated insulin delivery system includes the Bolus Priming System, a software automatically analyzing past continuous glucose monitoring values to trigger priming insulin bolus delivery isn the suspected presence of meal like glycemic disturbances
  FCL: The automated insulin delivery system does not include the Bolus Priming System, and therefore does not automatically command priming boluses.
Period: Overall Study
Arm/Group | Full Closed-loop (FCL) With Bolus Priming System (BPS) Followed by FCL Without BPS | Full Closed-loop (FCL) Without Bolus Priming System (BPS) Followed by FCL With BPS
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Closed-loop (FCL) With Bolus Priming System (BPS) Followed by FCL Without BPS | Full Closed-loop (FCL) Without Bolus Priming System (BPS) Followed by FCL With BPS | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (11.7) | 43.8 (14.9) | 38.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11
Baseline Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 6.3 (0.9) | 7.2 (1.3) | 6.7 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Daytime Percent Time-in-range
Description: Percentage of CGM values falling between 70 and 180 mg/dL during daytime (6am to midnight)
Time Frame: 18 hours
Measure: Mean (Standard Deviation); unit: percentage of CGM values
Groups:
- FCL With BPS: Fully closed-loop insulin delivery with bolus priming system
- FCL Without BPS: Fully closed-loop insulin delivery without BPS
Arm/Group | FCL With BPS | FCL Without BPS
Number analyzed (Participants) | 11 | 11
percentage of CGM values | 67.4 (15.1) | 65.1 (18.5)
Statistical Analysis 1: Comparison: FCL With BPS vs FCL Without BPS; Test type: Superiority; p = 0.4291, t-test, 2 sided; Mean Difference (Final Values) = 2.23, 95% CI 2-sided [-3.8 to 8.3], Standard Deviation 8.98

2. Secondary Outcome: Difference in Overall Percent Time-in-range
Description: Percentage of CGM values falling between 70 and 180 mg/dL
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: percentage of CGM values
Arm/Group | FCL With BPS | FCL Without BPS
Number analyzed (Participants) | 11 | 11
percentage of CGM values | 74.3 (13.6) | 73.1 (16.2)

3. Secondary Outcome: Difference in Daytime Percent Time-below-range
Description: Percentage of CGM values falling below 70mg/dL during daytime (6am to midnight)
Time Frame: 18 hours
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | FCL With BPS | FCL Without BPS
Number analyzed (Participants) | 11 | 11
percentage of CGM values | 0 [0 to 2.1] | 0 [0 to 1.3]

4. Secondary Outcome: Difference in Overall Percent Time-below-range
Description: Percentage of CGM values falling below 70mg/dL
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | FCL With BPS | FCL Without BPS
Number analyzed (Participants) | 11 | 11
percentage of CGM values | 0 [0 to 1.6] | 0 [0 to 1]

ADVERSE EVENTS:
Time Frame: From protocol entry through last study date which is approximately one month per participant
Description: Adverse Event definitions are the same as clinicaltrials.gov. Please see protocol for further details of adverse event reporting.
Groups:
- Full Closed-loop (FCL) With Bolus Priming System (BPS); Full Closed-loop (FCL) Without Bolus Priming System (BPS): Two separate 24-hour periods during where fully closed loop (FCL) control is used with & without the Bolus Priming system (BPS) active (BPS is designed to recognize meal ingestion & deliver a quick priming dose of insulin prior to extreme blood sugar excursions.) These will be separated by a 24-hour challenge period which will involve further meal & exercise challenges. During these 24-hour periods, participants will be followed for the experimental meals as part of the Study Controller Sessions to compare blood glucose control with & without the BPS. The study meals & activities will be standardized between study sessions.
  During a washout period, we will test the RocketAP system in FCL with further challenges:
  * A session of high-intensity interval training
  * A high-carbohydrate, high-fat meal
  * Ingestion of a bolus of simple sugar
  FCL+BPS: The automated insulin delivery system includes the Bolus Priming System, a software automatically analyzing past continuous glucose monitoring values to trigger priming insulin bolus delivery isn the suspected presence of meal like glycemic disturbances
  FCL: The automated insulin delivery system does not include the Bolus Priming System, and therefore does not automatically command priming boluses.
Arm/Group | Full Closed-loop (FCL) With Bolus Priming System (BPS) | Full Closed-loop (FCL) Without Bolus Priming System (BPS)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Closed-loop (FCL) With Bolus Priming System (BPS) (N=11) | Full Closed-loop (FCL) Without Bolus Priming System (BPS) (N=11)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) — Vomiting induced by exercise, not device-related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT05528770/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT05528770/ICF_001.pdf